CLINICAL TRIAL: NCT05706285
Title: Comparing Postoperative Analgesic Effects of Intrathecal Morphine With Erector Spina Plane Block in Open Gastrectomy Surgery
Brief Title: Comparing Intrathecal Morphine With Erector Spina Plane Block in Open Gastrectomy Surgery
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Beliz Bilgili, Associate Professor, Marmara University Pendik Training and Research Hospital
Other Study IDs: MarmaraUniv
Record Dates: First submitted 2023-01-04; First posted 2023-01-31 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Opioid Use; Post Operative Pain; Pain Assessment Scales
Keywords: erector spina plane block; intrathecal morphine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erector Spina Plane Block and Intravenous Patient Controlled Analgesia
  Interventions: Procedure: Regional Block Comparison
- Intrathecal Morphine and Intravenous Patient Controlled Analgesia
  Interventions: Procedure: Regional Block Comparison

INTERVENTIONS:
Procedure: Regional Block Comparison — Comparing postoperative pain and opioid consumption in groups

SUMMARY:
Open gastrectomy causes severe postoperative pain due to wide surgical incisions, retraction of the abdominal wall and direct manipulation of the visceral organs. It leads to delayed postoperative recovery, increased medical expenses and poor surgical outcomes. Epidural analgesia, intrathecal morphine and patient-controlled analgesia are frequently used in the postoperative pain management of abdominal surgeries. Intrathecal morphine is applied as a standard protocol in many centers due to its ease of application and effective pain control. However; it has undesirable effects such as postoperative nausea-vomiting, itching and most importantly respiratory depression. Regional interfascial plane blocks, such as erector spina plane block, have recently been popular in clinical practice to provide postoperative pain control. Erector spina plane block, when placed preoperatively, is expected to reduce opioid consumption and improve outcomes. The primary implication of this study is to compare postoperative pain scores and opioid consumption. It is also aimed to compare the effectiveness of Numeric Rating Scale and Clinically Aligned Pain Assessment Tool used in postoperative pain assesment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients undergoing open gastrectomy surgery

Exclusion Criteria:

* Patients with solid organ dysfunction
* Patients who receive opioid or corticosteroid medication prior to surgery
* Patients with bleeding diathesis
* Patients with psychiatric disorders
* Patients who can not be contacted after surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old undergoing open gastrectomy surgery in Marmara University Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessment with Numeric Rating Scale (NRS) | 48 hours
  In a Numerical Rating Scale (NRS), patients are asked to choose the number between 0 and 10, that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas ten represents 'the worst pain ever possible'
Postoperative pain assessment with Clinically Aligned Pain Assessment (CAPA) Tool | 48 hours
  CAPA tool functions as a conversation guide to gather categorical information during the course of a natural conversation. It focuses on how comfortable the patient is, whether discomfort is improving or worsening, whether the patient is able to participate in recovery activities and if pain is interfering with sleep.The clinician then codes and documents the conversation. Patient does not rate any scale or check boxes of responses.
Comparison of postoperative opioid consumption between two groups via Patient Controlled Analgesia (PCA) device | 48 hours
  Intravenous patient-controlled analgesia (PCA) is a system of opioid delivery that consists of an infusion pump interfaced with a timing device. Intravenous morphine consumption will be recorded via PCA device, then it will be documented in mg/kg units.

SECONDARY OUTCOMES:
Comparison of the frequency of treatment related complications | 48 hours
  Bradycardia, hypotension, sedation, respiratory depression, urinary retention, itching, need for rescue analgesics.
Participant satisfaction | 48 hours
  Whether the patient is very pleased/ satisfied/ unsatisfied/ complainant with the pain treatment will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided